CLINICAL TRIAL: NCT00382590
Title: A Randomized Phase II Study of the Combination of 5-Azacytidine With Valproic Acid (VPA) Versus Low-Dose Ara-C in Patients With AML/MDS Not Eligible for Other Studies
Brief Title: Azacytidine With Valproic Acid Versus Ara-C in Acute Myeloid Leukemia (AML)/ Myelodysplastic Syndrome (MDS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0177
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Myelodysplastic Syndrome; Leukemia; MDS; Azacytidine; 5-Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; Ara-C; Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Valproic Acid; VPA; Depakene
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Azacitidine; Cytarabine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-Aza + VPA (Active Comparator): 5-Azacytidine (5-Aza) 75 mg/m^2 subcutaneously daily + Valproic Acid (VPA) 50 mg/m^2 orally daily, each for 7 days
  Interventions: Drug: 5-Azacytidine; Drug: Valproic Acid (VPA)
- Ara-C (Active Comparator): Low-Dose Ara-C 20 mg twice daily subcutaneously for 10 days.
  Interventions: Drug: Ara-C

INTERVENTIONS:
Drug: 5-Azacytidine — 75 mg/m^2 daily for 7 days (days 1-7) via subcutaneous injection.
  Other Names: Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin
  Arms: 5-Aza + VPA
Drug: Ara-C — 20 mg twice daily via subcutaneous injection for 10 days.
  Other Names: Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
  Arms: Ara-C
Drug: Valproic Acid (VPA) — 50 mg/m^2 orally daily days 1-7.
  Other Names: VPA; Depakene
  Arms: 5-Aza + VPA

SUMMARY:
Primary Objective:

1. To evaluate whether 5 azacytidine (5-aza)/valproic acid (VPA) or low dose ara-C produces longer event free survival time in patients age > or = 60 years with untreated Acute Myeloid Leukemia (AML) or high risk Myelodysplastic Syndrome (MDS) who are typically ineligible for, or not placed on, studies of new agents.

Secondary Objective:

1. To evaluate whether pre-treatment methylation/acetylation status in AML/MDS blasts predicts response to either therapy or whether the ability of the 5 azacytidine + valproic acid combination to induce demethylation or acetylation parallels response.

DETAILED DESCRIPTION:
5-aza is a chemotherapy drug with activity in leukemia and MDS. Researchers hope that VPA will increase the effects of 5-aza. Low-dose Cytarabine (ara-C) is considered the standard of care for the treatment of leukemia and MDS in older patients not eligible for other therapies.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have blood drawn (about 2 teaspoons) for routine tests. You will also have a bone marrow biopsy and aspiration performed. To collect a bone marrow biopsy/aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive 5-aza and VPA. Participants in the other group will receive ara-C alone. At first, there will be an equal chance of being assigned to either group. As the study goes along, however, the chance of being assigned to the treatment that has worked best so far will increase.

Participants in the 5-aza and VPA group will receive 5-aza as an injection under the skin once a day for 7 days in a row. On these same 7 days, participants in this group will also take VPA by mouth twice a day or 3 times a day based on your weight. Seven (7) days is considered 1 treatment cycle. Both drugs will be taken at the same time. Cycles will be repeated every 4 to 6 weeks.

Participants in the ara-C group will receive ara-c twice a day as an injection under the skin for 10 days (1 cycle). Cycles will be repeated every 4 to 6 weeks.

You will be monitored with routine blood tests (about 1-2 teaspoons each time) 2-3 times a week during this study.

You may receive up to 12 cycles of therapy. You may be taken off study early if the disease gets worse or intolerable side effects occur.

Once you go off study, you will have standard follow-up as is required by your primary physician.

This is an investigational study. 5-aza is approved by the FDA for MDS. VPA is approved by the FDA for epilepsy. Their use together in this study is experimental. Ara-C is approved for acute myelogenous leukemia. About 70 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have untreated AML, or untreated MDS with > 10% blasts in marrow or blood.
2. They must be at least age 60.
3. They must either have a serum creatinine > 1.9 mg/ml, a serum bilirubin > 1.9 mg/ml, or a Zubrod performance status of 3 or 4.
4. Alternatively, they must not be candidates for protocols of higher priority.
5. They must provide written consent.

Exclusion Criteria:

1) Must not have the cytogenetic abnormalities inv (16), t (16;16) t (8;21), or t (15;17). The relatively good prognoses of patients with these findings do not warrant use of 5 azacytidine, + valproic acid or low-dose ara-C (LDAC).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 09/20/05 through 11/01/06. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Eleven (11) patients were registered, one (1) patient was not eligible and was taken off study prior to receiving study drug.
Groups:
- Ara-C: Low-Dose Cytarabine (Ara-C) 20 mg twice daily subcutaneously for 10 days.
Period: Overall Study
Arm/Group | 5-Aza + VPA | Ara-C
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-Aza + VPA | Ara-C | Total
Number analyzed (Participants) | 4 | 6 | 10
Age Continuous [Median (Full Range); unit: years] | 75 [70 to 79] | 76.5 [71 to 86] | 75.5 [70 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Patient response defined by: Death, Resistant to Therapy [no major hematologic improvement using International Myelodysplastic Syndromes (MDS) Working Group (Cheson B, Bennett J, Kantarjian H et al, Blood 2006) criteria after a maximum of 4 courses], or Relapse.
Time Frame: Evaluated every 3 weeks, following 4 courses (16/24 weeks ) and till study end
Population: The analysis was per intention to treat. One participant was inevaluable for response.
Measure: Number; unit: Participants
Arm/Group | 5-Aza + VPA | Ara-C
Number analyzed (Participants) | 4 | 5
Participants
  Death | 0 | 0
  Resistant to Therapy | 4 | 5
  Relapse | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year 2 months
Arm/Group | 5-Aza + VPA | Ara-C
Serious Adverse Events (participants affected / at risk) | 4/4 | 6/6
Other Adverse Events (participants affected / at risk) | 2/4 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Aza + VPA (N=4) | Ara-C (N=6)
Elevated liver function test (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Right periocular hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Left ocular hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lethargic fall (Nervous system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Atrail fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Aza + VPA (N=4) | Ara-C (N=6)
Arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (General disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
fatigue (Gastrointestinal disorders) | 0 (0) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
depression (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No